CLINICAL TRIAL: NCT02209987
Title: A Phase 1 Study to Evaluate the Absolute Bioavailability, Safety, and Tolerability of Subcutaneous GS-5745 in Healthy Subjects
Brief Title: Absolute Bioavailability, Safety, and Tolerability of Subcutaneous GS-5745 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-326-1430
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GS-5745 SC (Experimental): Participants will receive a single dose of GS-5745 by SC injection.
  Interventions: Drug: GS-5745 SC
- GS-5745 IV (Experimental): Participants will receive a single dose of GS-5745 by IV infusion.
  Interventions: Drug: GS-5745 IV

INTERVENTIONS:
Drug: GS-5745 SC — GS-5745 150 mg administered by SC injection formulated as a sterile, aqueous buffered solution in a single-use pre-filled syringe
  Arms: GS-5745 SC
Drug: GS-5745 IV — GS-5745 150 mg administered by IV infusion formulated as a sterile, aqueous buffered solution in single-use glass vials
  Arms: GS-5745 IV

SUMMARY:
This study will estimate the absolute bioavailability of subcutaneously injected GS-5745, characterize the safety, tolerability, and pharmacokinetics (PK) of GS-5745 after subcutaneous (SC) injection and intravenous (IV) administration, and evaluate the formation of anti-GS-5745 antibodies after SC and IV administration.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, individuals must be in good general health based upon medical history and physical examination
* Females, of childbearing potential, and males must agree to utilize protocol specific contraception methods
* Screening laboratory evaluations must be within defined thresholds

Exclusion Criteria:

* Infection with hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV)
* Pregnant and lactating females
* History of clinically significant illness (including psychiatric or cardiac) or any other medical disorder that may interfere with individual treatment and/or adherence to the protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
PK profile of GS-5745 | Predose and postdose on Days 1 and Day 11, and Weeks 2, 3, 4, 6, and 8
  This composite endpoint will measure the plasma PK profile of GS-5745. The following parameters will be measured, where applicable:
  * Cmax: maximum observed concentration of drug in plasma
  * AUClast: concentration of drug from time zero to the last quantifiable concentration
  * AUC0-inf: area under the plasma concentration versus time curve starting with time zero to infinity

SECONDARY OUTCOMES:
Incidences of adverse events and laboratory abnormalities | Up to 8 weeks
  This composite endpoint will measure the safety and tolerability profile of GS-5745.

CONTACTS AND LOCATIONS:
Overall Officials: Bittoo Kanwar, MD, Study Director — Gilead Sciences
Locations (1):
- Christchurch, New Zealand